CLINICAL TRIAL: NCT05592171
Title: A Randomized, Controlled, Open-label Study of the Safety and Efficacy of Occlusafe® Assisted Microwave Alone or in Combination With DEB-TACE Compared to Microwave in Combination With DEB-TACE in the Treatment of Intermediate Size HCC
Brief Title: Occlusafe® Assisted MW Alone or With DEB-TACE Compared to MW With DEB-TACE in the Treatment of HCC
Acronym: SEASON-HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Collaborators: A.O.U. Città della Salute e della Scienza (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Ospedaliera Universitaria Policlinico (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Terumo Europe N.V. (Industry); Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Laura Crocetti, Principal Investigator, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21704
Record Dates: First submitted 2022-10-17; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: HCC

STUDY DESIGN:
Intervention Model Description: Randomized open-label interventional study on a medical device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Occlusafe assisted MWA+ DEB-TACE (Other)
  Interventions: Procedure: Microwave ablation + Occlusafe + DEB-TACE
- Occlusafe assisted MWA (Other)
  Interventions: Procedure: Microwave ablation + Occlusafe
- MWA+ DEB-TACE (Other)
  Interventions: Procedure: Microwave ablation + DEB-TACE

INTERVENTIONS:
Procedure: Microwave ablation + Occlusafe + DEB-TACE — Microwave ablation (MW) is based on the production of heating by friction given by the oscillation of water molecules.
  After positioning and inflating the Occlusafe® balloon in the artery that connects to the HCC nodule, the blood flow tends to go preferentially to the HCC nodule compared to the healthy liver. The increase in the water content in the tumor area, after using the Occlusafe® balloon microcatheter, could increase the ability of microwave ablation to cover larger volumes in a shorter time.
  The delivery of drug-releasing microspheres (DEB-TACE) at the same time as microwave ablation, could promote the arrest of tumor growth.
  Arms: Occlusafe assisted MWA+ DEB-TACE
Procedure: Microwave ablation + Occlusafe — Microwave ablation (MW) is based on the production of heating by friction given by the oscillation of water molecules.
  After positioning and inflating the Occlusafe® balloon in the artery that connects to the HCC nodule, the blood flow tends to go preferentially to the HCC nodule compared to the healthy liver. The increase in the water content in the tumor area, after using the Occlusafe® balloon microcatheter, could increase the ability of microwave ablation to cover larger volumes in a shorter time.
  Arms: Occlusafe assisted MWA
Procedure: Microwave ablation + DEB-TACE — Microwave ablation (MW) is based on the production of heating by friction given by the oscillation of water molecules.
  The delivery of drug-releasing microspheres (DEB-TACE) at the same time as microwave ablation, could promote the arrest of tumor growth.
  Arms: MWA+ DEB-TACE

SUMMARY:
The goal of this Interventional Study is to compare the efficacy profile and safety of three treatments in patients with HCC nodule.

Patients will be randomly divided in three arms:

1. Occlusafe assisted MWA+ DEB-TACE
2. Occlusafe assisted MWA
3. MWA+ DEB-TACE

The primary objectives are evaluate the safety of the three treatments; evaluate the effectiveness of treatments one month after the procedure (defined as complete ablation of macroscopic tumor at one month of follow-up), verifying the possible superiority of arm 1 and arm 2 compared to arm 3.

The secondary objective is: time to local disease recurrence.

DETAILED DESCRIPTION:
Microwave ablation (MW) is based on the production of heating by friction given by the oscillation of water molecules.

The delivery of drug-releasing microspheres (DEB-TACE) at the same time as microwave ablation, could promote the arrest of tumor growth.

After positioning and inflating the Occlusafe® balloon in the artery that connects to the HCC nodule, the blood flow tends to go preferentially to the HCC nodule compared to the healthy liver. In addition, the flow is slowed down inside the nodule due to the drop in the resistance of the tumor arteries, resulting in stagnation of intranodular blood. The increase in the water content in the tumor area, after using the Occlusafe® balloon microcatheter, could increase the ability of microwave ablation to cover larger volumes in a shorter time.

In parallel, the delivery of drug-releasing microspheres (DEB-TACE) is provided both with inflation with Occlusafe® and without. This will allow to verify if a better treatment efficiency can be achieved in the peripheral ablation areas.

The study also includes a third control arm, consisting of ablation and DEB-TACE without Occlusafe®.

There is currently no interventional radiological treatment in the European guidelines to be preferred for HCC nodules 3-5cm in size in non-surgical patients.

Since these procedures are used in clinical practice, but the guidelines do not indicate a gold standard for non-surgical loco-regional treatment of HCC larger than 3 cm, the study aims to compare the efficacy profile and safety of the three treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age;
* any ethnicity;
* Patient with almost one HCC 3-5cm with biopsy according to EASL/EORTC guidelines;
* Patient is not candidate for liver resection;
* Child Pugh A;
* Eastern Cooperative Oncology Group (ECOG) performance status 0;
* Willing to sign an informed consent form, indicating awareness of the investigational nature of this study that is in keeping with the policies of the institution.

Exclusion Criteria:

* Have previously received therapeutic treatment for HCC outside the study protocol;
* Have extrahepatic metastasis;
* Have portal or hepatic vein tumor invasion/thrombosis;
* Baseline laboratories:

Platelet count < 50,000/mm3; INR > 1,5;

- Baseline Chemistry: Serum creatinine ≥ 2.0 mg/dL or calculated creatinine clearance (CrCl) ≤30.0 mL/min; Serum bilirubin > 3.0 mg/dL;

* Are pregnant or breast-feeding. In women of childbearing potential, a negative serum pregnancy test is required prior to study treatment;
* Have contraindications to receiving doxorubicin;
* Have other concurrent malignancy (subjects with treated squamous cell carcinoma of the skin or basal cell carcinoma of the skin may be included), evidence of extrahepatic cancer from their primary malignancy, or ongoing, medically significant active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-10-17 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CIRSE classification of complications | immediately after the procedure
  Evaluate the safety of the three treatments by CIRSE classification
Number of Participants With Treatment-Related Adverse Events as Assessed by CIRSE classification of complications | 30 days
  Evaluate the safety of the three treatments by CIRSE classification
Number of participants with complete response according to mRECIST one month after the procedure | one month
  Number of participants with complete response according to mRECIST one month after the procedure, verifying the possible superiority of arm 1 and arm 2 compared to arm 3.

SECONDARY OUTCOMES:
Time to local disease recurrence | 1 month, 4 months, 7 months, 10 months, 13 months
  ● Relapse-free survival analysis. Appearance of local disease recurrence on CT examination with contrast medium performed according to the scheduled timing

CONTACTS AND LOCATIONS:
Overall Officials: Laura Crocetti, MD, PhD, Principal Investigator — University of Pisa
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, Italy